CLINICAL TRIAL: NCT06560528
Title: Clinical Study on the Efficacy and Safety of Disitamab Vedotin Combined With Tislelizumab and Capecitabine in the Perioperative Treatment of Locally Advanced Gastric Cancer With HER2 Overexpression
Brief Title: Disitamab Vedotin Combined With Tislelizumab and Capecitabine in the Perioperative Treatment of Locally Advanced Gastric Cancer With HER2 Overexpression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20241606
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: RC48-ADC; HER2
MeSH Terms: conditions — Stomach Neoplasms | interventions — disitamab vedotin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination with Disitamab Vedotin and with Tislelizumab and Capecitabine (Experimental): Subjects will receive Disitamab Vedotin combined with Tislelizumab and Capecitabine for 3 cycles (Q3W) in the neoadjuvant phase and 5 cycles (Q3W) of treatment in the adjuvant phase.
  Disitamab Vedotin：2.5 mg/kg，Q3W； Tislelizumab：200 mg，Q3W； Capecitabine：1000 mg /m2, PO, bid d1-14, Q3W.
  Interventions: Drug: combination with Disitamab Vedotin and with Tislelizumab and Capecitabine

INTERVENTIONS:
Drug: combination with Disitamab Vedotin and with Tislelizumab and Capecitabine — Subjects will receive Disitamab Vedotin combined with Tislelizumab and Capecitabine for 3 cycles (Q3W) in the neoadjuvant phase and 5 cycles (Q3W) of treatment in the adjuvant phase.
  1. Disitamab Vedotin：2.5 mg/kg，Q3W；
  2. Tislelizumab：200 mg，Q3W；
  3. Capecitabine：1000 mg /m2, PO, bid d1-14, Q3W.

SUMMARY:
The efficacy and safety of combination with Disitamab Vedotin and with Tislelizumab and Capecitabine for perioperative treatment of locally advanced gastric cancer with HER2 overexpression.

DETAILED DESCRIPTION:
This study included 40 patients with HER2 overexpression in locally advanced gastric cancer or gastroesophageal junction adenocarcinoma, who received treatment with Disitamab Vedotin combined with Tislelizumab and Capecitabine. The patient has not received any previous anti-tumor systemic therapy. HER2 expression is defined as immunohistochemistry (IHC) as 2+or 3+. Subjects who meet the inclusion criteria but do not meet the exclusion criteria will receive perioperative treatment after enrollment. Perioperative treatment includes neoadjuvant therapy and adjuvant therapy.

Subjects will receive Disitamab Vedotin combined with Tislelizumab and Capecitabine for 3 cycles in the neoadjuvant phase and 5 cycles of treatment in the adjuvant phase.

ELIGIBILITY:
Inclusion Criteria:

* 1) Volunteer to take part in the study ;
* 2) Age 18~75 (including 75), male or female;
* 3) Gastric cancer or adenocarcinoma of gastroesophageal junction confirmed by histology and/or cytology;
* 4) Clinical stage Ⅱ, Ⅲ (cT2-4a ,N+ or -, M0, AJCC 8th);
* 5) Have not received systematic treatment;
* 6) The HER2 immunohistochemistry (IHC) test result is IHC 3+or 2+, and the previous test results of the subject (confirmed by the investigator) are acceptable;
* 7) At least one assessable lesion (RECIST 1.1 );
* 8) Expected survival time ≥ 6 months;
* 9) ECOG 0-1;
* 10) Major organs are functioning normally；

Exclusion Criteria:

* 1) Have a history of malignant tumors other than gastric cancer, except for the following two cases:

  1. The patient has received possible curative treatment and there is no evidence of the disease within 5 years;
  2. The resected skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ and other carcinoma in situ were successfully received;
* 2) Suffering from diseases that affect the absorption, distribution, metabolism or clearance of the study drug (such as severe vomiting, chronic diarrhea, intestinal obstruction, absorption disorder, etc.);
* 3) Have received allogeneic stem cells or solid organ transplantation in the past;
* 4) Patients who have received other anti-tumor systemic therapy in the past (including traditional Chinese medicine with anti-tumor indications), and have been less than 4 weeks from the completion of treatment to the administration of this study, or the adverse events caused by previous treatment have not recovered to ≤ CTCAE level 1 (except hair loss and pigmentation);
* 5) Previous or current congenital or acquired immunodeficiency disease;
* 6) Active or previously recorded autoimmune diseases or inflammatory diseases (including but not limited to: autoimmune hepatitis, interstitial pneumonia, inflammatory bowel disease, systemic lupus erythematosus, vasculitis, uveitis, hypophysitis, hyperthyroidism or hypothyroidism, asthma requiring bronchodilators, etc.), vitiligo or asthma that has completely alleviated in childhood, Those who do not need any intervention after adulthood can be included;
* 7) Systemic immunosuppressive drugs were used within 2 weeks before enrollment, or were expected to be required during the study, except for the following:

  1. Corticosteroids for intranasal, inhalation, external or local injection (such as intra-articular injection);
  2. The dose of prednisone or other equivalent systemic corticosteroids does not exceed 10 mg/day;
  3. Preventive use of corticosteroids for hypersensitivity;
* 8) Allergic to the study drug;
* 9) Thrombosis or thromboembolism events occurred in the past 6 months, such as stroke and/or transient ischemic attack, deep vein thrombosis, pulmonary embolism, etc;
* 10) Patients at risk for severe bleeding；
* 11) Cardiovascular diseases with significant clinical significance;
* 12) Other significant clinical and laboratory abnormalities, which the researchers think affect the safety evaluation;
* 13) Serious infection in active period or poorly controlled clinically;
* 14) Not recovered from the operation;
* 15) Pregnant or lactating women, and women or men with fertility who are unwilling or unable to take effective contraceptive measures;
* 16) Other situations that the investigator thinks are not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete remission rate (PCR) | up to 1 years
  Pathological complete response (pCR) rate is defined as the proportion of participants whose tumor in the stomach and lymph node completely disappeared, as determined by a pathologist.

SECONDARY OUTCOMES:
Objective response rate(ORR) | up to 3 years
  Overall response rate ( ORR) is defined as proportion of participants who have a best response of CR or PR
Major pathological response rate (MPR) | up to 1 year
  Major pathological response (MPR) rate is defined as the proportion of participants whose percentage of residual tumor in the stomach and lymph node decreased to < 10%, as determined by a pathologist
1-3-years event-free survival rate of 3year (EFS) | up to 3 years
  1-3 years event-free survival (EFS) rate is defined as proportion of participants who have no event, including disease progression, cessation of treatment for any reason, or death after 1-3 years of radical treatment.
1-3 years overall survival (OS) rate | up to 3 years
  1-3 years overall survival (OS) rate is defined as proportion of participants who survived 1-3 years after radical treatment
Adverse Events（AEs） | up to 3 years
  Defined as the proportion of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Han Liang, Ph.D, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; Xuewei Ding, Ph.D, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (2):
- China (2):
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Xuewei Ding, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No